CLINICAL TRIAL: NCT04191460
Title: Guided by Light: Optimizing Surgical Excision of Oral Cancer Using Real-time Fluorescence Imaging
Brief Title: Fluorescence-guided Surgery Using cRGD-ZW800-1 in Oral Cancer
Acronym: GuidedbyLight
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Stijn Keereweer, Principal Investigator, Erasmus Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 12175; 2019-003416-30 (EudraCT Number)
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck; Oral Cancer; Squamous Cell Carcinoma of the Oral Cavity
Keywords: cRGD-ZW800-1; fluorescence-guided surgery; image-guided surgery; fluorescence imaging; cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- WP-I dose A (Experimental): n=7. Injection of 0.05 mg/kg cRGD-ZW800-1, within 16-20 hours before imaging/surgery
  Interventions: Drug: cRGD-ZW800-1.
- WP-I dose B (Experimental): n=7. Injection of (to be determined) mg/kg RGD-ZW800-1, within (to be determined) hours before imaging/surgery.
  Interventions: Drug: cRGD-ZW800-1.
- WP-II selected dose (Experimental): n=14: expansion cohort (n=14) will be added to the group of patients that had received the selected dose in WP-I. Injection of 0.05 ór (to be determined) mg/kg cRGD-ZW800-1, within 48 hours before imaging/surgery.
  Interventions: Drug: cRGD-ZW800-1.

INTERVENTIONS:
Drug: cRGD-ZW800-1. — Injection of cRGD-ZW800-1 within 48 hours before imaging/surgery

SUMMARY:
This is a two-staged clinical trial to investigate the feasibility of intraoperative Fluorescence Imaging (FLI) to adequately assess tumor margins in patients with oral cancer using cRGD-ZW800-1.

DETAILED DESCRIPTION:
Work package I:

In WP-I, the preferred dose of the agent for imaging of margins in oral cancer will be determined. The signal-to-noise ratio will be determined in dose group A (n=7), which will receive 0.05 mg/kg of the tracer, 16-20 hours before surgery. After an interim evaluation of this ratio, the second dose group B (n=7) will receive either a higher or a lower dosage (to be determined) of the tracer. After inclusion of all patients (n=14), the dose with the highest intraoperative signal-to-noise ratio will be selected.

Work package II:

In WP-II, an expansion cohort (n=14) will be added to the group of patients that had received the selected dose in WP-I. In this group of 21 patients, it will be determined if FLI can improve the rate of adequate surgical resection margins. As secondary research questions, the following aspects will be assessed:

* sensitivity, specificity, positive and negative predictive values of FLI;
* colocalization with immunohistochemistry;
* change in surgical management; incremental operation time;
* FLI of excised cervical lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with biopsy-proven squamous cell carcinoma of the oral cavity, eligible for surgical resection of the primary tumor;
2. ≥ 18 years of age;
3. Before patient registration, written informed consent must be given according to ICH/GCP, and national/local regulations;
4. Screening ECG and clinical laboratory test results are within normal limits, or if any are outside of normal limits they are considered to be clinically insignificant.

Exclusion Criteria:

1. Previous surgery, chemotherapy or radiotherapy to the oral cavity;
2. History of a clinically significant allergy or anaphylactic reactions to any of the components of the agent.
3. Patients pregnant or breastfeeding, lack of effective contraception in male or female patients with reproductive potential;
4. Patients with renal insufficiency (eGFR<60);
5. Patients with a previous kidney transplantation in the medical history;
6. Immuno-compromised patients who do not have the ability to respond normally to an infection due to an impaired on weakened immune system, caused by either a pre-existing disease or concomitant medications;
7. Any condition that the investigator considers to be potentially jeopardizing the patient's well-being or the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
WP-I: (Highest) mean tumor-to-background ratio (TBR) | up to 48 ours post-dose
  Two dosages of cRGD-ZW800-1 are tested in two groups of each 7 patients. An expansion cohort (n=14) will be added to the dose group that yields the highest TBR.
WP-II: Rate of adequate (i.e. >5mm clear) tumor resection margins. | through histopathology, up to max 4 weeks post-op

SECONDARY OUTCOMES:
WP-II: Sensitivity, specificity, positive and negative predictive values | through histopathology, up to max 4 weeks post-op
WP-II: Co-localization of FLI with immunohistochemistry on pathology slides | through histopathology, up to max 4 weeks post-op
WP-II: Percentage of extra tissue resection based on FLI-driven frozen sections | through histopathology, up to max 4 weeks post-op
WP-II: Operation time | through histopathology, up to max 4 weeks post-op
WP-II: FLI of lymph node metastases after neck dissection | through histopathology, up to max 4 weeks post-op

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus University Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: First in-human study of cRGD-ZW800-1 in patients with colorectal cancer — https://pubmed.ncbi.nlm.nih.gov/32345649/